CLINICAL TRIAL: NCT06668545
Title: Immunohistochemical Analysis of CD 71 Levels in the Placenta of Preeclamptic and Normotensive Pregnancies and Comparison With Neonatal Outcomes
Brief Title: Investigating CD 71 in Preeclamptic Pregnancies
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: MCBU_Preeklampsi
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Preeclampsia; Placenta Diseases
Keywords: Preeclampsia; inos; enos; cd71
MeSH Terms: conditions — Pre-Eclampsia; Placenta Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Biospecimen Retention: Samples With DNA — placenta tissues and umlical cord tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:: Patients with preeclampsia
- Group 2:: Patients without preeclampsia

SUMMARY:
Objective: Upon reviewing studies aimed at understanding and investigating the pathogenesis of preeclampsia, it has been observed that CD71 has not been previously examined. Therefore, the increase in CD71 is associated with placental dysfunction and mechanisms affecting fetal growth restriction. The exact pathogenesis of CD71, which is known to play a role in such mechanisms, has not been fully understood. Consequently, this study may contribute to understanding and elucidating the development of preeclampsia. This study aims to investigate the levels of CD71 and NOS in the placentas of pregnant women with high and normal blood pressure and to compare these findings with neonatal outcomes.

Method: This prospective randomized controlled study will be conducted at the Department of Obstetrics and Gynecology, Manisa Celal Bayar University, involving patients diagnosed with preeclampsia. The planned sample size was calculated using the G power 3.1.9.7 program, with an effect size of 1.153, 95% power, and a 0.5% type I error rate. The calculated sample size for the case group is 39 and for the control group is also 39. When the planned sample size is reached, sample collection will be terminated, and histopathological examinations will be conducted.

Study Group: Patients with preeclampsia Control Group: Patients without preeclampsia

During the hospitalization of the preeclampsia patients for delivery, after clamping of the umbilical cord following the birth of the baby (after the connection between mother and baby has ceased), a 2 ml (one teaspoon) blood sample will be taken from the cord blood, centrifuged, and the serum sample will be separated and stored at -80 degrees Celsius. In the post-delivery process, a 3x3 cm piece will be taken from the umbilical cord, which will be disposed of as medical waste, and from the placenta (the baby's afterbirth), encompassing all layers. The collected tissue samples will be preserved in a container with 10% formalin. At the time of sample collection, both the cord blood and placenta samples will be in a waste state, ensuring that there is no connection left between the mother and baby, thus eliminating any risk of harm to either during the sampling process. The tissues (placenta, umbilical cord) and the 2 ml (one teaspoon) blood sample from the umbilical cord will be collected, centrifuged, and the serum sample separated, to be stored at -80 degrees Celsius for future similar studies and projects.

Preeclampsia is a serious complication during pregnancy that poses potential risks to both the mother and the baby. Early diagnosis and appropriate management can reduce complications and safeguard maternal-fetal health. Biomarkers of preeclampsia play a significant role in the understanding and management of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy under 37 weeks
* Age range 18-50
* Being literate in Turkish
* Not having any additional disease
* Agreeing to participate in the study

Exclusion Criteria:

* High-risk pregnancies (gestational hypertension, preeclampsia, HELLP syndrome, chronic hypertension, gestational and pregestational diabetes, cholestasis, intrauterine growth retardation, etc.)
* Multiple pregnancy
* Pregnant women under the age of 18
* Smoking
* Medication use (excluding routinely used food supplements during pregnancy)
* Additional disease (thyroid, renal failure, liver failure, hepatitis, heart disease, connective tissue disease, etc.)
* Immunosuppressive use
* Presence of active or chronic infection
* Presence of active or chronic inflammatory disease
* Patients who gave birth at an external center or later chose to withdraw from the study
* Patients who did not have any exclusion criteria at the time of Preeclampsi or when blood was drawn for the control group, but who later developed any exclusion criteria.
* Premature birth of patients included in the control group

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Preeclampsi Patients
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
2% women's with PPROM placenta tissues and umblical cord while birth. Placenta tissues and umblical cord Staining will be Measured by inos,enos,cd71 immunohistochemistry | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Kemal Sarsmaz, Manisa, Yunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes